CLINICAL TRIAL: NCT04106752
Title: Timing of Meal and Caffeine Intake on Substrate Use and Exercise Efficiency in Healthy Individuals
Brief Title: Timing of Meal and Caffeine Intake on Substrate Use and Exercise Efficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: NUT.EF.01
Record Dates: First submitted 2019-09-12; First posted 2019-09-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-01

CONDITIONS: Healthy
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- meal followed by caffeine (Active Comparator): A standardized meal consisting of 2 slices of toast bread, organic peanut butter and jam was given to the participant. One and a half hours later, the participant ingested a caffeinated drink (3 mg per kg body weight of caffeine powder dissolved in water). After 30 mins, resting EE was measured using FM for 15 min while seated on the comfortable seat, and then for 5 min while seated on a cycle ergometer. Participants were then asked to pedal at 60 revolutions per minute (rpm) for 5 min per load at 20 watts (W), 35W, 50W, 65W, 80 W respectively. During cycling, EE was being measured using the FM, HR was monitored and rating of perceived exertion (RPE) was recorded in the last minute of every load cycle.
  Interventions: Dietary Supplement: Caffeine
- Caffeine followed by meal (Active Comparator): Caffeine was given to the participant. After 1.5 hours the standardized meal was given followed by the same protocol mentioned above.
  Interventions: Dietary Supplement: Caffeine
- caffeine only (Active Comparator): Caffeine will be given to the participant. 2 hours later the same protocol mentioned above will be applied
  Interventions: Dietary Supplement: Caffeine
- Meal only (Active Comparator): A standardized meal will be given to the participant. 2 hours later the same protocol mentioned above will be applied.
  Interventions: Dietary Supplement: Caffeine
- meal plus caffeine (Active Comparator): A standardized meal + a caffeinated drink (3 mg/kg of body weight of caffeine powder dissolved in water) will be given to the participant. 2 hours later resting EE is measured using a facemask (FM) for 10 min while seated on a cycle ergometer . The participant will be asked to pedal at 60 revolutions per minute (rpm) for 5 min per load at 20 watts (W), 35W, 50W, 65W, 80 W respectively.
  Interventions: Dietary Supplement: Caffeine

INTERVENTIONS:
Dietary Supplement: Caffeine — Provide caffeine supplements with or without meal before exercise

SUMMARY:
During the past decades, considerable emphasis has been directed to analyzing the potential role of caffeine on substrate use and exercise performance. Research shows that caffeine ingestion prior to exercise has beneficial effects on submaximal exercise capacity and time trial protocols. This effect is mediated by an increase in plasma free fatty acids and intramuscular triglyceride utilization, preserving muscle and liver glycogen. Generally, a dose between 4 - 9 mg/kg body mass is administered to athletes in order to observe a positive or ergogenic effect. Caffeine ingestion (6 mg/kg) improved exercise performance in a long duration protocol (2 hours + ~ 30 min time trial) regardless of the administration time (1 hour before or during exercise). Lower doses of caffeine (~ 1.5 mg/kg), when added to a carbohydrate solution increased exercise performance in a similar fashion. In rats, caffeine has been shown to have a biphasic action on postprandial glucose metabolism. When ingested before a meal, hepatic glycogenesis is blunted. Its ingestion during and after a meal allows glycogenesis to occur. Manipulating meal and caffeine timing before low intensity exercise, comparable to every-day life activities, is of great interest in assessing substrate use and muscular efficiency. it would be also interesting to see how this meal or caffeine timing manipulation influence the energetics of different phenotypes.

DETAILED DESCRIPTION:
Research shows that caffeine ingestion prior to exercise has beneficial effects on moderate to high exercise performance. Generally, a dose between 4 - 9 mg/kg body mass is administered to athletes in order to observe a positive effect.

The aims of the study are the following: first, to investigate the effect of caffeine and/or meal on energy supply (% from fat and carbohydrate) during low intensity exercise. Second, to investigate the effect of timing and order of the above on energy supply before, during, and after exercise. Lastly, to assess exercise efficiency following the above protocols (work accomplished relative to the calories spent to accomplish the work).

Healthy, untrained male and female subjects will be recruited for this study. Subjects will be excluded if they had a previous history of any limitation on physical ability, cardiovascular disease, taking supplements or medicine that might affect their metabolic rate, claustrophobic, or unstable bodyweight during the past 6 months. Subjects will be defined as sedentary, with a maximum of 30 minutes of moderate physical activity per day (assessed by questionnaire) excluding daily activities.

During the first visit, participants will be informed about the experiment protocol, if agreed, they should give a written consent, answer a questionnaire (lifestyle), and get anthropometric and body composition measurements.

On the day of testing, subjects will come to the laboratory at 08:00 fasted. All participants will be requested to avoid physical activity, caffeine, and dietary supplements in the 24h prior to testing.

Energy expenditure is measured by indirect calorimetry. Briefly, participants will sit in a comfortable seat, using a ventilated hood with baseline energy expenditure. During this period, the participant is instructed to relax and avoid movements. Heart rate monitoring is included using a heart rate belt. Participants then complete the following protocols on five separate days (separated by at least 48 hours) in a randomized order:

Protocol 1:

A standardized meal (2 slices of toast bread + butter + Jam ~ 500 kcal) + caffeine (~200 mg) will be given to the participant. 2 hours later resting energy expenditure is measured using a facemask for 10 min while seated on a cycle ergometer. The participant will be asked to pedal at 60 revolutions per minute for 5 min per load at 20 watts (W), 35W, 50W, 65W, 80 W respectively.

Protocol 2:

A standardized meal will be given to the participant. 2 hours later caffeine will be given followed by the same protocol mentioned above.

Protocol 3:

Caffeine will be given to the participant. 2 hours later a standardized meal will be given followed by the same protocol mentioned above.

Protocol 4:

Caffeine will be given to the participant. 2 hours later the same protocol mentioned above will be applied.

Protocol 5:

A standardized meal will be given to the participant. 2 hours later the same protocol mentioned above will be applied.

Manipulating meal and caffeine timing before low intensity exercise, comparable to every-day life activities, is of great interest in assessing energy supply and muscular efficiency in humans.

There is no risks related to the study. Exercise is maintained at a low-to-moderate level comparable to everyday life. All data related to the subjects will be coded (# and initials, i.e. A001_ELIFAR) and kept confidential.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female individual between 18 and 30 years old,
* normal weight or overweight

Exclusion Criteria:

* Subjects will be excluded if they are not covered by (University health insurance) HIP,
* subjects with the previous history of any limitation on physical ability,
* Subjects with cardiovascular disease,
* Subjects taking supplements or medicine that might affect their metabolic rate,
* claustrophobic,
* Subjects with unstable body weight during the past 6 months.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-29 (Actual)

PRIMARY OUTCOMES:
Changes in respiratory quotion | 24 months
  Compare respiratory quotient (RQ) values (indicator of the substrate being used) during low level exercise after caffeine and/or meal intake
Exercise efficiency | 24 months
  Calculate exercise efficiency (delta work/ delta energy) during different protocols. The more efficient the participant is the more work he or she can do with the same amount of energy

CONTACTS AND LOCATIONS:
Overall Officials: Elie-Jacques Fares, PhD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No